CLINICAL TRIAL: NCT01740349
Title: EVALUATION OF THE PILLCAM™ COLON CAPSULE ENDOSCOPY (PCCE) IN PEDIATRIC ULCERATIVE COLITIS
Brief Title: Evaluation Of The Pillcam™ Colon Capsule Endoscopy (Pcce-2) In Pediatric Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, EVALUATION OF THE PILLCAM™ COLON CAPSULE ENDOSCOPY (PCCE) IN PEDIATRIC ULCERATIVE COLITIS, Azienda Policlinico Umberto I
Other Study IDs: PCCE-2 GIVEN
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2012-11

CONDITIONS: Pediatrics, Colon Capsule Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 30 children with UC: This prospective pilot study of 30 pediatric subjects, that are indicated for standard colonoscopy due to follow-up of ulcerative colitis (UC), examines the Given Diagnostic System and the PillCam Colon Capsule in comparison to standard colonoscopy.

SUMMARY:
This prospective pilot study of 30 pediatric subjects, that are indicated for standard colonoscopy due to follow-up of ulcerative colitis (UC), examines the Given Diagnostic System and the PillCam Colon Capsule in comparison to standard colonoscopy.

This study aims

1. To evaluate and compare the accuracy of PillCam ™ Colon capsule endoscopy (PCCE) with standard colonoscopy in the evaluation of colon in pediatric ulcerative colitis.
2. To evaluate the safety of PillCam ™ Colon capsule endoscopy (PCCE) in pediatric age.

ELIGIBILITY:
ELIGIBILITY Ages Eligible for Study: 6-18 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Inclusion criteria:

Subjects must meet one the following inclusion criteria to be eligible for enrollment into this proposed study:

* diagnosis of UC made at least 3 months before the enrolment;
* subject was referred for standard colonoscopy and endoscopic follow-up in Ulcerative colitis
* signed informed consent. Exclusion criteria

The presence of any of the following will exclude a subject from study enrollment:

* Subject has dysphagia
* Subject has renal insufficiency
* Subject is known or suspected structuring CD.
* Subject has a cardiac pacemaker or other implanted electro medical devices.
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, a swallowable device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the Given® Diagnostic System include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure. This prospective pilot study will evaluate the performance of PCCE in visualizing the colon of children with UC. All subjects to be enrolled will be appropriate candidates for standard colonoscopy based on their clinical indication.
  Each subject will undergo PCCE. PCCE results will be compared with that of a colonoscopy procedure.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the accuracy of PillCam ™ Colon capsule endoscopy (PCCE) with standard colonoscopy in the evaluation of colon in pediatric ulcerative colitis. | Day 3 (after colonoscopy and CCE-2)
  Accuracy parameters (sensitivity, specificity, NPV, PPV) of PCCE compared to standard colonoscopy in pediatric Ulcerative Colitis.

SECONDARY OUTCOMES:
To evaluate the safety of PillCam ™ Colon capsule endoscopy (PCCE) in pediatric age. | Day 3 (after colonoscopy and CCE-2)
  Number, type and severity of adverse events with both PCCE and standard colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza - University of Rome, Rome, Italy, Italy

REFERENCES:
- [Derived] Oliva S, Di Nardo G, Hassan C, Spada C, Aloi M, Ferrari F, Redler A, Costamagna G, Cucchiara S. Second-generation colon capsule endoscopy vs. colonoscopy in pediatric ulcerative colitis: a pilot study. Endoscopy. 2014 Jun;46(6):485-92. doi: 10.1055/s-0034-1365413. Epub 2014 Apr 28. PMID 24777427